CLINICAL TRIAL: NCT00906984
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere® For Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: TheraSphere® for Treatment of Unresectable Hepatocellular Carcinoma
Acronym: TheraSphere
Status: Approved for marketing | Type: Expanded Access
Sponsor: University of California, Irvine (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Nadine Abi-Jaoudeh, Professor of Clinical Radiology, University of California, Irvine
Other Study IDs: 20022242; CA60396 (Other Grant/Funding Number: National Cancer Institute); UCI 01-61 (Other: CFCCC)
Record Dates: First submitted 2007-12-27; First posted 2009-05-21 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasm; Primary Liver Cancer
Keywords: Hepatocellular carcinoma; Liver cancer; Primary liver cancer; Unresectable liver cancer; Unresectable hepatocellular carcinoma; TheraSphere
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Device: TheraSphere — Given IV

SUMMARY:
The purpose of this protocol is to provide TheraSphere treatment for patients with liver cancer who cannot be treated by surgery. The effect on the tumor and any side effects of TheraSphere treatment will be examined. This study will provide supervised and limited access to TheraSphere treatment at University California Irvine Medical Center.

TheraSphere is a medical device containing yttrium-90 (Y-90), a radioactive material that has been used previously in the treatment of liver tumors. When Y-90 is incorporated into very tiny glass beads (TheraSphere), it can be injected to the liver through blood vessels supplying the liver. This allows a large dose of radiation to be delivered to the tumor with less risk of toxic effects from radiation to other parts of the body or to healthy liver tissue. The radiation from TheraSphere is contained within the body and becomes minimally active within 7 days after treatment due to physical decay. The glass beads remain in the body, but do not cause any health problems. TheraSphere has been approved for use in the treatment of liver cancer in the United States by the Food and Drug Administration on a limited basis.

DETAILED DESCRIPTION:
This protocol provides TheraSphere treatment for patients with liver cancer who cannot be treated by surgery. Patients with hepatocellular carcinoma will be evaluated for eligibility for this treatment with the following: physical examination, medical history, blood tests requiring approximately 2 tablespoons of blood, EKG, CT or MR of chest to examine lungs, CT or magnetic resonance (MR) of abdomen to evaluate liver, stomach and intestines, and bone scan to rule out spread of disease to bones. If eligible on initial screening, patients will proceed to a second stage of screening, including an hepatic angiogram to confirm treatment can be provided safely and to highlight the blood vessels supplying the liver, and a nuclear medicine study (Tc-99m MAA scan) to display the blood flow to the lungs, stomach and intestines.

When it is determined treatment can be delivered safely, patients will receive TheraSphere via the hepatic artery through blood vessels supplying the liver on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of intrahepatic carcinoma. The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers such as Alpha-fetoprotein assay (AFP) (clinical diagnosis).
* The cancer must be unresectable.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score 0 - 2
* Age ≥ 18 years.
* Able to comprehend and read the study information sheet in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Any pre-treatment laboratory findings within 15 days of treatment demonstrating:

  * Absolute granulocyte count ≤ 1,500/ul
  * Platelet count ≤ 75,000/μl
  * Serum creatinine ≥ 2.0 mg/dl
  * Serum bilirubin ≥ 2.0 mg/dl
* Any of the following contraindications to angiography and selective visceral catheterization:

  * History of severe allergy or intolerance to any contrast media, narcotics, sedatives, or atropine
  * Bleeding diathesis, not correctable by usual forms of therapy
  * Severe peripheral vascular disease that would preclude catheterization.
* Portal hypertension with portal venous shunt away from the liver.
* Evidence of potential delivery of greater than 16.5 millicurie (mCi) (30 Gy absorbed dose) of radiation to the lungs on either: 1) first TheraSphere administration; or 2) cumulative delivery of radiation to the lungs > 30 Gy over multiple treatments.
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow.
* Significant extrahepatic disease representing an imminent life-threatening outcome.
* Severe liver dysfunction or pulmonary insufficiency.
* Active uncontrolled infection.
* Significant underlying medical or psychiatric illness.
* Pregnant women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, MD, Principal Investigator — University of California, Irvine
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- [Background] Salem R, Thurston KG. Radioembolization with 90Yttrium microspheres: a state-of-the-art brachytherapy treatment for primary and secondary liver malignancies. Part 1: Technical and methodologic considerations. J Vasc Interv Radiol. 2006 Aug;17(8):1251-78. doi: 10.1097/01.RVI.0000233785.75257.9A. PMID 16923973
- [Background] Salem R, Thurston KG. Radioembolization with 90yttrium microspheres: a state-of-the-art brachytherapy treatment for primary and secondary liver malignancies. Part 2: special topics. J Vasc Interv Radiol. 2006 Sep;17(9):1425-39. doi: 10.1097/01.RVI.0000235779.88652.53. PMID 16990462
- [Background] Salem R, Thurston KG. Radioembolization with yttrium-90 microspheres: a state-of-the-art brachytherapy treatment for primary and secondary liver malignancies: part 3: comprehensive literature review and future direction. J Vasc Interv Radiol. 2006 Oct;17(10):1571-93. doi: 10.1097/01.RVI.0000236744.34720.73. PMID 17056999
- See also: More information on TheraSphere — http://www.therasphere.com